CLINICAL TRIAL: NCT01894971
Title: The Effect of Thermal Damage of Ligasure® to Destroy Cornual Portion of Fallopian Tube Tissue
Brief Title: The Effect of Ligasure® to Destroy Cornual Portion of Fallopian Tube
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Joong Kim, Assistant Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-06-25
Record Dates: First submitted 2013-06-25; First posted 2013-07-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Recruiting; Completed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- twice coagulated side of fallopian tube (Experimental): twice coagulated side of fallopian tube once coagulated sied of fallopian tube
  Interventions: Device: The Effect of Ligasure® to Destroy Cornual Portion of Fallopian Tube

INTERVENTIONS:
Device: The Effect of Ligasure® to Destroy Cornual Portion of Fallopian Tube

SUMMARY:
Single-center prospective randomized trial to evaluate the effect of thermal damage of Ligasure® to destroy cornual portion of fallopian tube tisse.

Right of Left side of fallpian tube is randomized and coagulated one more time than other side before cut off. The pathologist evaluate the amount of fallopian tube tissue left at both cornual portion of cut off specimen.

DETAILED DESCRIPTION:
When investigators perform salpingectomy, both side of cornual portion of the uterus are coagulated by Ligasure®. The randomized, the same word selected side of the fallopian tube is coagulated one more time at the cornual portion than unselected other side of fallopian tube. Hypothesis is that the side selected and coagulated twice would have less fallopian tube tisse left at fianl pathology than the side only once coagulated by Ligasure®.

ELIGIBILITY:
Inclusion Criteria:

* female 35-50
* premenopausal
* plan to perform hysterectomy

Exclusion Criteria:

* disease in fallopian tube before surgery
* has history of pelvic inflammatory disease

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Remnant fallopian tube tissue after coagulation wiht Ligasure® | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Tae Joong Kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Unable to connect to PubMed to validate , last attempt on June 25, 2013 at 11:11 AM EDT